CLINICAL TRIAL: NCT05598463
Title: The Effect of AR-based Home Rehabilitation Exercise Combined With Wearable Sensor (IMU) on Physical Function, Depression, Physical Activity, and Self-efficacy in the Elderly: A Exploratory Study on the Effectiveness of OASIS Pro
Brief Title: The Exploratory Study of AR-based Home Rehabilitation Exercise Combined With Wearable Sensor (IMU) in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Korea Medical Device Development Fund grant (Unknown)
Responsible Party: Principal Investigator, JiHye Hwang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OASIS Pro_study
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Telerehabilitation; Geriatrics; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented reality and wearable sensor-based home rehabilitation exercise (Experimental): Experimental group performs augmented reality and wearable sensor-based home rehabilitation exercise for 4 weeks. And then, their exercise compliance is monitored by medical staff.
  Interventions: Device: OASIS Pro
- Control group (No Intervention): Control group is asked to maintain their own physical activity amount, not involve the regular exercise program additionally for 4 weeks after enrollment.

INTERVENTIONS:
Device: OASIS Pro — This device can track the joint movement and provide real-time feedback on the exercise performance and accuracy using Kinect camera sensor, and Wearable sensor (IMU). This device is connected to the website, which available for medical staff prescribe the exercise protocol and monitor individual exercise adherence.
  Arms: Augmented reality and wearable sensor-based home rehabilitation exercise

SUMMARY:
According to the results of a systematic literature review and meta-analysis based on recent studies on exercise interventions for the elderly based on augmented reality, virtual reality, and functional games, these technology-based exercise interventions It was confirmed that there was a positive effect on the function. In addition, it was found to indirectly enhance the motivation for performing physical exercise. In a recent similar study, when an exercise program was applied to 27 elderly people for 3 months through an exercise device that can measure body movements in real time through a Kinect camera, the physical activity of the elderly was induced, and the sustainability of exercise was increased. It is expected that this will be effective in preventing muscle loss in the elderly.

However, due to the limitations of the existing Kinect camera, motions that have to be performed lying down or when exercising while wearing black clothes overlapped the movements of the lower extremities and caused motions in which the joint position could not be accurately tracked, thereby reducing the accuracy of exercise performance. There were limitations that could not be measured. In order to solve these technical limitations and improve clinical applicability, several existing studies have conducted inertia measurement that can accurately detect the motion of lower extremity joints by measuring the speed, acceleration, and direction of body movement in the X, Y, and Z axes. I started using Inertial Measurement Units (IMUs). Wearable sensors such as IMUs can enhance motor learning by providing immediate feedback on motor performance and motor errors. In addition, in the case of commercial camera systems such as the Kinect camera, if the user's appearance is obscured by other objects, there is a disadvantage that it is not detected. This is an important advantage in a home environment where there is no medical supervision, and this risk can be minimized, especially for the elderly who are at risk of falling. Previously, several literatures have applied the IMU sensor to the elderly and patients with total knee/hip arthroplasty and confirmed the effect.

In this study, the OASIS Pro to be used can receive visual feedback by applying a virtual environment (number of exercises, exercise target point, and holding time) with the real home environment as the background. The Kinect camera can be used alone, and at the same time, an IMU sensor can be attached to the lower extremities to perform precise movements. The user performs the exercise prescribed by the manager (medical staff), and when the exercise is finished, the user can receive feedback on the accuracy and performance. Administrators can create and manage individual exercise protocols through OASIS-Manager. Therefore, the investigators intend to prove the effectiveness of OASIS Pro by applying augmented reality-based home rehabilitation exercise combined with IMU sensor to the elderly and confirming the effect on physical ability, depression, physical activity, and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Seniors over 65

Exclusion Criteria:

1. Persons with severe comorbidities that make exercise impossible due to unstable angina, acute myocarditis, aneurysm, uncontrolled cardiovascular disorder, etc.
2. Those with neurological and visual impairments to the extent that movement is difficult
3. Those with dizziness during exercise
4. Those who participate in a regular exercise program more than twice a week or are receiving physical therapy
5. Those who have difficulty in communicating and maintaining necessary education and maintenance in the research process
6. Others who should not perform exercise as judged by a medical professional

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of Short Physical Performance Battery (SPPB) | Enrollment, 1month
  comparison between groups in change of SPPB score between baseline (enrollment) and after 1 months.
  This max score is 12 (range from zero to 12), meaning higher score, and higher physical performance.

SECONDARY OUTCOMES:
Change of Exercise Self-efficacy | Enrollment, 1month, 2 month
  This consists of 9 items, and scale ranges from zero (not sure at all) to 10 (very sure), representing the higher score, and higher exercise self-efficacy.
Change of depression (using Short form of Geriatric depression scale, SGDS-K) | Enrollment, 1month, 2 month
  A total of 15 questions, marked with yes or no. It is a scale of 15 points, and the higher the score, the higher the depression.
Change of physical activity (using Korean Version of Physical Activity Scale for the Elderly, K-PASE) | Enrollment, 1month, 2 month
  The possible score range is from 0 to 360, with higher scores indicating more physical activity.

OTHER OUTCOMES:
Satisfaction with Intervention device (OASIS Pro) | 1month
  It consists of multiple-choice questions about overall satisfaction with OASIS Pro and usefulness, and subjective-type questions about satisfaction and improvements.
  minimum and maximum values have 0 and 5 points respectively. Higher scores mean better outcome.
Usability with Intervention device (OASIS Pro) | 1month
  It is evaluated by System Usability Scale (SUS), comprises of the 10 items. Higher score represents the higher usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No